CLINICAL TRIAL: NCT02102841
Title: Investigating the Role of Skin Resident T Cells in Atopic Eczema and Responses to Antigen Challenge
Brief Title: Investigating Immune Mechanisms in Atopic Eczema
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment no longer feasible
Sponsor: University College, London (Other)
Collaborators: Dermatrust (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13/0410; 14/LO/0243 (Other: Health Research Authority)
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Skin biopsy (Experimental): 5mm skin punch biopsy on forearm
  Interventions: Procedure: Skin biopsy
- Skin suction blister (Experimental): Skin suction blister induced on forearm
  Interventions: Procedure: Skin suction blister
- Mantoux, skin biopsy, suction blister (Experimental): 0.1ml tuberculin purified protein derivative (PPD) is injected intradermally into an area of non-lesional skin on the volar aspect of each of the patient's forearms. This is followed by a skin biopsy on one arm and induction of a skin suction blister on the other arm.
  Interventions: Procedure: Skin biopsy; Procedure: Skin suction blister; Biological: Mantoux test

INTERVENTIONS:
Procedure: Skin biopsy
  Arms: Mantoux, skin biopsy, suction blister; Skin biopsy
Procedure: Skin suction blister
  Arms: Mantoux, skin biopsy, suction blister; Skin suction blister
Biological: Mantoux test
  Other Names: Tuberculin PPD (SSI)
  Arms: Mantoux, skin biopsy, suction blister

SUMMARY:
The aim of this study is to investigate the mechanisms behind the immune dysfunction that occurs in atopic eczema (or atopic dermatitis).

DETAILED DESCRIPTION:
Atopic eczema is a chronic inflammatory skin disease that affects 15-20% of children and 12% of adults and leads to significant loss of quality of life. It results from a complex interaction of genetic and environmental factors, and is characterised by dysregulation of the cutaneous immune system. Specifically, in the skin of eczema patients there is a persistence of T lymphocytes (a crucial cell involved in regulating the immune system), and an overproduction of certain cytokines (signalling molecules that are essential in producing inflammatory responses).

The study intends to investigate the causes of atopic eczema by examining the number, characteristics and function of T lymphocytes in the skin and the blood of eczema patients, as well as the types of cytokine they produce. To achieve this the investigators aim to take skin biopsies, tissue fluid (from induced skin suction blisters) and blood samples from adult eczema patients and healthy controls for analysis. Additionally, in these groups a cutaneous immune response will be initiated by injecting tuberculin protein purified derivative (the Mantoux test) into the skin, to further investigate how the behaviour of T lymphocytes varies between eczema patients and healthy controls.

This research is important in view of the high prevalence of atopic eczema in the population. An improved understanding of its causes will hopefully lead to more effective treatments for this condition in future.

ELIGIBILITY:
Inclusion Criteria:

* History of atopic dermatitis (according to United Kingdom Working Party's diagnostic criteria)
* Previous Bacillus Calmette-Guerin vaccination

Exclusion Criteria:

* Unable to give written informed consent
* Previous history of hypersensitivity to local anaesthetic (for skin biopsy) or tuberculin PPD (for skin test)
* Pregnancy or breast feeding
* History of tuberculosis
* Recent infection or immunisation (within last month)
* Known immunodeficiency e.g. HIV infection, primary immunodeficiency, any history of chemotherapy or radiotherapy
* Systemic steroids within the last month or any other immunosuppressive medications (eg. methotrexate, ciclosporin or azathioprine) within the previous 3 months
* Phototherapy within the previous 28 days
* Treatment with potent topical corticosteroids or tacrolimus ointment within the previous 7 days
* Significant co-morbidity (diabetes, renal failure, liver failure, heart failure)
* On warfarin or known bleeding disorder
* History of neoplasm in last 10 years (not including basal cell carcinoma)
* Previous keloid scarring

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Number of regulatory T cells in lesional skin of atopic dermatitis patients compared to healthy volunteers | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Rustin, MBBS MRCP MD, Principal Investigator — Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free London NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Williams HC, Burney PG, Hay RJ, Archer CB, Shipley MJ, Hunter JJ, Bingham EA, Finlay AY, Pembroke AC, Graham-Brown RA, et al. The U.K. Working Party's Diagnostic Criteria for Atopic Dermatitis. I. Derivation of a minimum set of discriminators for atopic dermatitis. Br J Dermatol. 1994 Sep;131(3):383-96. doi: 10.1111/j.1365-2133.1994.tb08530.x. PMID 7918015